CLINICAL TRIAL: NCT01484925
Title: Notch Signaling and Novel Biomarkers for Barretts Esophagus
Brief Title: BETERNet Notch Signaling and Novel Biomarkers for Barretts Esophagus
Status: Completed | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 22211
Record Dates: First submitted 2011-12-01; First posted 2011-12-05 (Estimated); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: Barrett's Esophagus
Keywords: Barrett's esophagus
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- With Barrett's Esophagus: Patients who have been diagnosed in the past with Barrett's Esophagus
- Without Barrett's Esophagus: Patients without Barrett's Esophagus will be asked to take part so that comparison can be made with patients' tissue for those with the condition and those without the condition.

SUMMARY:
This research study hopes to identify new molecular markers in the tissue of Barrett's esophagus that will help physicians better understand and manage this condition. Patients undergoing an upper endoscopy will be asked to complete a gastroesophageal reflux disease (GERD) questionnaire, provide a blood sample and allow additional biopsies to be taken during the procedure.

DETAILED DESCRIPTION:
This research study hopes to identify new molecular markers in the tissue of Barrett's esophagus that will help physicians better understand and manage this condition. Currently there is very little understanding as to how Barrett's esophagus develops and why some people with Barrett's esophagus go on to develop esophageal cancer. The purpose of this study is to develop a better understanding of how these processes occur. The investigators also hope to use the information from this study to identify new molecular markers that the investigators can use to better determine who will or will not go on to develop esophageal cancer. Patients who have been diagnosed in the past with Barrett's esophagus will be asked to participate. Patients without Barrett's esophagus will be asked to take part so that the investigators can compare tissue from patients without the conditions to those with the conditions.

ELIGIBILITY:
Inclusion Criteria:

For BE patients:

* History of histologically confirmed BE, defined as endoscopically-suspected BE with intestinal metaplasia with globlet cells on esophageal biopsies,
* BE length C1M1 or C0M2
* Age 18 years

Exclusion Criteria:

* History of gastric or esophageal surgery
* Inability to give informed consent
* Erosive esophagitis seen on upper endoscopy
* History of prior endoscopic therapy for BE 5 (for controls) History of intestinal metaplasia on previous esophageal, GE junction or cardia biopsies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Barretts Esophagus with and without associated dysplasia or cancer and controls with and without gastro-esophageal reflux.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2011-11; Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Falk, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center, Philadelphia, Pennsylvania, United States